CLINICAL TRIAL: NCT02333318
Title: A Single Ascending Dose Escalation Clinical Trial to Investigate Safety and Pharmacokinetics of VVZ-149 Injection in Healthy Older Male Volunteers
Brief Title: A Single Ascending Dose Escalation to Investigate Safety and PK of VVZ-149 Injection in Healthy Older Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vivozon, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: PT-VVZ149-02
Record Dates: First submitted 2014-12-24; First posted 2015-01-07 (Estimated); Last update posted 2019-03-13 (Actual); Status verified 2015-01

CONDITIONS: Healthy
MeSH Terms: interventions — Water; Injections

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Single Dose_VVZ-149 injection (Experimental): 1. Cohort A (50-64 years old), Cohort B (65-84 years old)
  2. For 2.5, 5mg/kg
  3. 4-hr intravenous infusion of VVZ-149 injection
  4. 6 subjects will be administered within each age group. Total 24 subjects will participate.
  Interventions: Drug: VVZ-149 injection
- Loading/Maintenance_VVZ-149 injection (Experimental): 1. Cohort A (50-64 years old) This trial is conducted only in the Cohort A one week after the single IV infusion.
  2. For Loading + Maintenance dose: 0.75 mg/kg+ 0.55 mg/kg/h, 1.5 mg/kg + 1.10 mg/kg/h
  3. intravenous infusion
  4. 4 subjects will be randomly assigned within each dose group, respectively. Total 8 subjects will participate.
  Interventions: Drug: VVZ-149 injection
- Loading/Maintenance_Placebo (Placebo Comparator): 1. Cohort A (50-64 years old)
  2. For Loading + Maintenance dose: 0.75 mg/kg+ 0.55 mg/kg/h, 1.5 mg/kg + 1.10 mg/kg/h
  3. intravenous infusion
  4. 2 subjects will be randomly assigned within each dose group, respectively. Total 4 subjects will participate.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: VVZ-149 injection — Colorless, transparent liquid in water for injection
  Other Names: VVZ-149 injection or water for injection
  Arms: Loading/Maintenance_VVZ-149 injection; Single Dose_VVZ-149 injection
Other: Placebo — water for injection
  Other Names: VVZ-149 injection or water for injection
  Arms: Loading/Maintenance_Placebo

SUMMARY:
The objective of this study is to investigate the safety, tolerability and pharmacokinetics (PK) of VVZ-149 injection after a single dose or loading/maintenance dose in healthy older male volunteers.

DETAILED DESCRIPTION:
VVZ-149 injection, an investigational product (IP) in this clinical study, is a multi-target analgesic drug candidate against glycine transporter type II (GlyT2) and serotonin receptor 2A (5HT2A). The target receptors have been known to play important roles in the induction and transmission of pain signals in the pain-related neural system. There have been efforts to develop new drugs that selectively antagonize the GlyT2 or 5HT2A, but it was unsuccessful due to limitations of single-target drugs. VVZ-149 showed morphine-comparable analgesic and gabapentin-comparable anti-allodynic effects in various rat models of pain.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who voluntarily agree to participate and sign an IRB-approved informed consent form (ICF) prior to receiving any of the screening procedures
2. Healthy male subjects aged between 50-84, inclusive at screening (the subjects aged 65 years or over can participate only in the single dose trial)
3. Subjects with body weights between 50-90 kg, inclusive and with body mass index (BMI) between 18.0-29.9 kg/m2, inclusive
4. Healthy subjects satisfying eligibility at screening (medical histories, physical examination, vital sign, electrocardiogram (ECG), hematology, clinical chemistry and urinalysis)
5. Subjects who willing to use an medicinal allowed method of contraception or sterility during the study period

Exclusion Criteria:

1. Subjects who have a presence or history of clinically significant hepatic, renal, neurologic, immunologic, pulmonary, endocrine, hematological, neoplastic, cardiovascular or psychiatric (e.g. mood disorders or obsessive-compulsive disorder) diseases (subjects with currently well-controlled conditions including hypertension, hyperlipidemia, arthritis, prostatic hypertrophy and cataracts may allow to participate at the discretion of the investigator.)
2. Subjects with chronic infection or meaningful acute infection
3. Subjects who have a history of clinically significant hypersensitivities or hypersensitivities to the ingredient of same family with IP and other drug (e.g. aspirin and antibiotics)
4. Subjects who have a family history of chronic pain or with a first-degree relative with chronic pain
5. Subjects who have a clinically significant ECG abnormalities or QTc interval >450 ms
6. Subjects who meet the following criteria at screening:

   * AST or ALT level > 3 times the upper limit of the normal range
   * Calculated eGFR by MDRD equation < 60 ml/min
   * Platelets ≤ 75,000/mm3, Hemoglobin ≤ 9 g/dL, Neutrophils absolute ≤ 1000/mm3
7. Subjects who show the following vital signs at the screening:

   * Systolic Blood Pressure (SBP): <92 mmHg or >160 mmHg
   * Diastolic Blood Pressure (DBP): <50 mmHg or >95 mmHg
8. Subjects who have a history of drug abuse or a positive urine screening for drug abuse
9. Subjects who have taken any prescribed or herbal medicine within one week before the first administration of the IP or any non-prescribed medicine or vitamin supplement within three days before the first administration of the IP (if all other conditions are satisfied, these subjects may be eligible for the trial as judged by the investigator)
10. Subjects who have participated in any other clinical trial within two months before the first administration of the IP
11. Subjects who have donated a unit of whole blood within two months or blood components within one month before the first administration of the IP, or who have received blood transfusion within one month before the first administration of the IP
12. Subjects who consume more than 21 units of alcohol per week (1 unit = 10 g of pure alcohol) or who are unable to abstain from drinking throughout the trial
13. Smokers who consume more than average of 10 cigarettes per day over the past three months or who are unable to abstain from smoking throughout the trial
14. Subjects who consume or are unable to abstain from products containing caffeine (e.g. coffee, green tea, black tea and sodas) within 24 hours before the first administration of the IP and until discharge from the hospital
15. Subjects judged ineligible for the study by the investigator for reasons of medical, psychological, social and geographical conditions causing poor study compliance

Ages: 50 Years to 85 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2014-07; Primary Completion 2014-09 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicity and maximum tolerated dose | 8 day
  Any Common Toxicity Criteria for Adverse Effects grade 3 or more adverse event , All significant toxicity judged by the investigator

SECONDARY OUTCOMES:
Safety and Tolerability as measured by Adverse event, physical examination, vital signs, 12-lead ECG, consecutive ECG, SpO2 monitoring and Clinical laboratory. | 8 day
  Adverse event, physical examination, vital signs, 12-lead ECG, consecutive ECG, SpO2 monitoring, Clinical laboratory

OTHER OUTCOMES:
The pharmacokinetics parameters: AUClast, AUCinf and Cmax | [Single Dose Trial] * Blood sampling (17 times) pre-dose and 0.25, 0.5, 1, 2, 3, 4, 4.25, 4.5, 5, 5.5, 6, 7, 8, 12, 24 and 32 h post-dose * Urine collection (5 times) pre-dose and 0-6, 6-12, 12-24 and 24-32 h post-dose [Loading/maintenance Dose Trial] *
  Blood sampling and urine sampling

CONTACTS AND LOCATIONS:
Overall Officials: Jae Yong Chung, MD, PhD, Principal Investigator — Seoul National University Bundang Hospital